CLINICAL TRIAL: NCT02725515
Title: A Randomized, Double-Blinded, Placebo-Controlled Study of the Effect of XmAb®5871 on Systemic Lupus Erythematosus Disease Activity
Brief Title: A Study of the Effect of XmAb®5871 in Patients With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Collaborators: PPD Development, LP (Industry); ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XmAb5871-04
Record Dates: First submitted 2016-01-08; First posted 2016-04-01 (Estimated); Results first posted 2019-08-09 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: Randomized (1:1, no stratification), Double-Blinded, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- XmAb5871 (Experimental): XmAb5871 administered by IV infusion for up to a total of 16 infusions
  Interventions: Biological: XmAb5871
- Placebo (Placebo Comparator): Placebo to match XmA5871 administered by IV infusion for up to a total of 16 infusions
  Interventions: Biological: Placebo to match XmAb5871

INTERVENTIONS:
Biological: XmAb5871
  Arms: XmAb5871
Biological: Placebo to match XmAb5871
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the ability of XmAb5871 to maintain Systemic Lupus Erythematosus (SLE) disease activity improvement achieved by a brief course of disease-suppressing steroid therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of SLE as defined by the ACR criteria
* Patients have a history of a (+) ANA, (+) ENA or a (+) anti-dsDNA serology documented within one year prior to randomization
* Investigator has assessed the patient and in their judgment, the SLE disease activity is not organ threatening
* Both investigator and patient agree that it is acceptable to discontinue their current immunosuppressant SLE medications and receive a brief course of IM steroid therapy
* If patients are on oral steroids, they must be on the equivalent of ≤15 mg/day of prednisone to enter screening, and must be able to taper to ≤10 mg/day by randomization

Exclusion Criteria:

* History or evidence of a clinically unstable/uncontrolled disorder, condition or disease, other than SLE that, in the opinion of the investigator would pose a risk to patient safety or interfere with the study evaluation, procedures or completion
* Patients who have organ threatening manifestations of SLE including active Class 3 or 4 lupus nephritis requiring induction or maintenance therapy or any other disorder for which stopping SLE therapy is contraindicated
* Active CNS lupus such as seizures or psychosis that in the opinion of the investigator would preclude participation
* Unstable hemolytic anemia or thrombocytopenia
* Patient is pregnant or breast feeding, or planning to become pregnant while participating in the study
* Use of any biologic therapy (including belimumab) within 6 months of randomization, or prior exposure to a monoclonal antibody directed to CD20 (such as rituximab) within 12 months of randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - UC San Diego, La Jolla, California
  - Loma Linda University, Loma Linda, California
  - East Bay Rheumatology Medical Group, San Leandro, California
  - Yale University School of Medicine, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Center For Rheumatology, Fort Lauderdale, Florida
  - Piedmont Atlanta Rheumatology, Atlanta, Georgia
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Joshua P June, DO, Lansing, Michigan
  - Washington University, St Louis, Missouri
  - Suny Downstate Medical Center, Brooklyn, New York
  - Feinstein Institute for Medical Research, Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Columbia University Medical Center, The Bronx, New York
  - CTRC University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - DJL Clinical Research, Charlotte, North Carolina
  - Paramount Medical Research and Consulting LLC, Cleveland, Ohio
  - Arthritis & Rheumatology Center of Oklahoma, PLLC, Oklahoma City, Oklahoma
  - Oklahoma Center for Arthritis Therapy & Research, Tulsa, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bombardier C, Gladman DD, Urowitz MB, Caron D, Chang CH. Derivation of the SLEDAI. A disease activity index for lupus patients. The Committee on Prognosis Studies in SLE. Arthritis Rheum. 1992 Jun;35(6):630-40. doi: 10.1002/art.1780350606. PMID 1599520
- [Background] Gladman DD, Ibanez D, Urowitz MB. Systemic lupus erythematosus disease activity index 2000. J Rheumatol. 2002 Feb;29(2):288-91. PMID 11838846
- [Derived] Merrill JT, Guthridge J, Smith M, June J, Koumpouras F, Machua W, Askanase A, Khosroshahi A, Sheikh SZ, Rathi G, Burington B, Foster P, Matijevic M, Arora S, Wang X, Gao M, Wax S, James JA, Zack DJ. Obexelimab in Systemic Lupus Erythematosus With Exploration of Response Based on Gene Pathway Co-Expression Patterns: A Double-Blind, Randomized, Placebo-Controlled, Phase 2 Trial. Arthritis Rheumatol. 2023 Dec;75(12):2185-2194. doi: 10.1002/art.42652. PMID 37459248

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First informed consent date: 16FEB2016 First randomization date: 07MAR2016 Last informed consent date: 09NOV2017 Last randomization date: 07DEC2017
Pre-assignment Details: After obtaining informed consent, IM depomedrol was administered and screening studies were performed over the 2-4 week screening period. Immunosuppressive therapy must have been stopped or tapered off by randomization on Day 1. Patients who did not meet the disease activity improvement criteria during the screening period were not randomized.
Period: Overall Study
Arm/Group | XmAb5871 | Placebo
Started | 53 | 52
Completed | 28 | 17
Not Completed | 25 | 35
Not completed — Refused infusion (no study treatment) | 1 | 0
Not completed — Loss of Improvement per Protocol | 14 | 25
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Non-Compliance With Study Drug | 0 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 7 | 2
Not completed — No Documented Disease Improvement | 0 | 1
Not completed — Completed Study Under Original Protocol | 0 | 1
Not completed — Lack of Response | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) Population: All patients who have received at least a partial dose of XmAb5871 or placebo. One patient was randomized to XmAb5871 but was never treated and withdrew from the study. This one patient is excluded from this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | XmAb5871 | Placebo | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Continuous [Median (Full Range); unit: years] | 45.5 [23 to 65] | 43.5 [20 to 64] | 45.0 [20 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 49 | 99
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 46 | 48 | 94
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 25 | 51
  White | 19 | 25 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 52 | 52 | 104
SLEDAI Total Score at Screening--Efficacy Evaluable Population [Median (Full Range); unit: units on a scale] — The Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) total score ranges between 0 and 105. The higher the score, the more significant is the degree of disease activity. Scores of 6 and above are considered to be consistent with active disease requiring therapy. Population: Efficacy Evaluable Population: All patients who:
  * Complete study through Day 225 assessments
  * Discontinue due to reaching the protocol specified LOI endpoint (and have not missed 2 or more consecutive doses prior to the LOI visit)
  * Discontinue due to drug-related adverse event (nonresponder)
  units on a scale
    number analyzed (Participants) | 50 | 42 | 92
    (all) | 8.0 [4 to 16] | 10.0 [2 to 18] | 10.0 [2 to 18]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Without Loss of Systemic Lupus Erythematosus Disease Activity Improvement on Day 225
Description: Landmark proportion of patients without loss of systemic lupus erythematosus disease activity improvement on Day 225
Time Frame: Day 225
Population: Efficacy Evaluable Population: All patients who:
  * Complete study through Day 225 assessments
  * Discontinue due to reaching the protocol specified LOI endpoint (and have not missed 2 or more consecutive doses prior to the LOI visit)
  * Discontinue due to drug-related adverse event (nonresponder)
Measure: Count of Participants; unit: Participants
Arm/Group | XmAb5871 | Placebo
Number analyzed (Participants) | 50 | 42
Participants | 21 | 12
Statistical Analysis 1: Comparison: XmAb5871 vs Placebo; Test type: Superiority; p = 0.1830, Barnard's Unconditional Exact Test P-val; Risk Difference (RD) = 13.4, 95% CI 2-sided [-6.6 to 32.6]

2. Secondary Outcome: Percentage of Patients Without Loss of Systemic Lupus Erythematosus Disease Activity Improvement on Day 169
Description: Landmark proportion of patients without loss of systemic lupus erythematosus disease activity improvement on Day 169
Time Frame: Day 169
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XmAb5871 | Placebo
Number analyzed (Participants) | 50 | 42
Participants | 29 | 17
Statistical Analysis 1: Comparison: XmAb5871 vs Placebo; Test type: Superiority; p = 0.1075, Barnard's Unconditional Exact Test P-val; Risk Difference (RD) = 17.5, 95% CI 2-sided [-3.7 to 37.3]

3. Secondary Outcome: Time to Loss of Systemic Lupus Erythematosus Disease Activity Improvement Achieved by a Short Period of IM Steroid Therapy in SLE Patients
Description: Loss of improvement was defined as worsening of disease activity that in the opinion of the principal investigator requires a change in treatment (exclusive of a decrease in oral steroids) AND one of:
  1. SELENA- SLEDAI increase of >=4 points from maximal improvement OR
  2. Worsening of at least 1 BILAG A or B score OR
  3. New BILAG A or B score.
Time Frame: From the date of randomization until the date of loss of Systemic Lupus Erythematosus Disease Activity Improvement, or the date of the final efficacy assessment, up to 239 days.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | XmAb5871 | Placebo
Number analyzed (Participants) | 50 | 42
days | 230 [197.0 to 239.0] | 131 [85.0 to 225.0]
Statistical Analysis 1: Comparison: XmAb5871 vs Placebo; Test type: Superiority; p = 0.0252, Log Rank; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.30 to 0.92]

ADVERSE EVENTS:
Time Frame: Adverse event summaries include events reported between randomization and the end of study visit (Day 253)
Description: Adverse events were reported by study center investigators using an electronic data capture system.
  Safety Population: All patients who have received at least a partial dose of XmAb5871 or placebo.
  One patient was randomized to XmAb5871 but was never treated and withdrew from the study. This one patient is excluded from adverse event summaries.
Arm/Group | XmAb5871 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 7/52 | 4/52
Other Adverse Events (participants affected / at risk) | 41/52 | 28/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XmAb5871 (N=52) | Placebo (N=52)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 1
Migraine (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | XmAb5871 (N=52) | Placebo (N=52)
Nausea (Gastrointestinal disorders) | 20 | 9
Headache (Nervous system disorders) | 12 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 6
Vomiting (Gastrointestinal disorders) | 9 | 1
Dizziness (Nervous system disorders) | 8 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 4
Urinary tract infection (Infections and infestations) | 5 | 3
Flushing (Vascular disorders) | 7 | 0
Nasopharyngitis (Infections and infestations) | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2
Acute sinusitis (Infections and infestations) | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Bronchitis (Infections and infestations) | 2 | 3
Hot flush (Vascular disorders) | 4 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 2
Peripheral swelling (General disorders) | 3 | 2
Anxiety (Psychiatric disorders) | 3 | 1
Fatigue (General disorders) | 4 | 0
Non-cardiac chest pain (General disorders) | 4 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Migraine (Nervous system disorders) | 3 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Tachycardia (Cardiac disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
Prior to database lock, an evaluation of early discontinuation rates indicated that the efficacy-evaluable population might be insufficient to power the primary analysis. An additional 15 patients were enrolled beyond the originally planned 90.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-07-29): https://cdn.clinicaltrials.gov/large-docs/15/NCT02725515/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/15/NCT02725515/SAP_001.pdf